CLINICAL TRIAL: NCT02369432
Title: Exploratory Study of the Cutaneous Penetration of Biodegradable Polymeric Microparticles in Atopic Dermatitis
Acronym: MicroIskin
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Difficulties in enrolling patients
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: University of Franche-Comté (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: API/2012/32
Record Dates: First submitted 2015-02-16; First posted 2015-02-24 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Atopic Dermatitis
Keywords: Drug carriers; Polymeric microparticles; Preferential accumulation in inflamed skin; Atopic dermatitis; Pilosebaceous follicles; Selective drug delivery; Drug reservoir
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group of healthy volunteers and group of patients (Experimental): * Healthy volunteers: Microparticles will be applied to the skin of the forearm and then a skin biopsy of this area will be performed
  * Patients suffering from atopic dermatitis: Microparticles will be applied to the skin of the forearm both to an area affected by dermatitis and to an area deprived from the disease. A skin biopsy of these two areas will be performed
  Interventions: Drug: Biodegradable and biocompatible polymeric microparticles containing a fluorochrome applied to the skin followed by a skin biopsy

INTERVENTIONS:
Drug: Biodegradable and biocompatible polymeric microparticles containing a fluorochrome applied to the skin followed by a skin biopsy

SUMMARY:
This proof of concept study aims to assess in patients suffering from atopic dermatitis if polymeric microparticles reach the pilosebaceous follicles of inflamed skin.

DETAILED DESCRIPTION:
Current treatments of inflammatory skin disorders such as acne, psoriasis or atopic dermatitis are primarily topical. They have the advantage of allowing the administration of active substances directly to the skin lesions.

However local treatments may have drawbacks (complex application, local and/or systemic side effects...) and cause poor compliance.

The use of drug carriers is viewed as one of the most promising strategies to target and control the release of active substances to various skin sites. Polymeric microparticles have shown to have a better stability and a more sustained release pattern than other types of drug vehicles such as liposomes.

Based on the results obtained in our preclinical experiments, this proof of concept study aims to assess, in patients suffering from atopic dermatitis, if biodegradable polymeric microparticles reach the pilosebaceous follicles of inflamed skin which would in turn serve as a reservoir of active substance.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers:

  * Volunteers over 18
  * Male volunteers under 65 or women of childbearing age (with a negative pregnancy test obtained at least 3 weeks before inclusion)
  * Caucasian volunteers
  * Volunteers having never shown any type of skin lesions regardless of its origin especially any allergic skin reactions.
  * Volunteers having signed a free and informed consent form
  * Volunteers affiliated to a social security system
* Patients:

  * Patients over 18
  * Male patients under 65 or women of childbearing age (with a negative pregnancy test obtained at least 3 weeks before inclusion)
  * Caucasian patients
  * Acute phase of atopic dermatitis with a SCORAD between 15 and 40
  * Patients suffering from atopic dermatitis skin lesions ≥ 1.5 cm² on the inside of the forearm
  * Patients having been treated by class II dermocorticoids with a two-week wash-out prior to inclusion
  * Patients having signed a free and informed consent form
  * Patients affiliated to a social security system

Exclusion Criteria:

* Participants under 18
* Pregnant or Breastfeeding women
* Post-menopausal women
* Patients having skin lesions adjacent to the selected area
* Patients with complications of atopic dermatitis
* SCORAD <15 or >40
* Patients being treated with a topical or a systemic treatment influencing the skin penetration of the microparticles
* Patients allergics to any component of the formulation
* Patients using cosmetic products on their forearms
* Patients planning to expose themselves to the sun
* Patients with a known immune deficiency
* Patients allergic to any product or device used before, during or after the skin biopsy
* Patients suffering from known wound healing disorders
* Patients with known inherited ou acquired hemostasis disorders
* Patients unable to follow the protocol requirements
* Patients currently involved in another clinical trial (or whose participation has ended less than 2 weeks before inclusion)
* Patients who are not affiliated to a social security system
* Patients in an exclusion period following participation in another clinical trial
* Incapacitated adults
* Participants placed under tutorship or curatorship
* Participants under judicial protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-02-20 (Actual); Primary Completion 2017-10-03 (Actual); Study Completion 2017-10-03 (Actual)

PRIMARY OUTCOMES:
Assessment of the penetration beyond the stratum corneum in human skin (fluorochrome contained in the particle will be detected by confocal microscopy) | Day 3
  * Healthy volunteers: Microparticles are applied to the skin of the forearm and then a skin biopsy of this area is performed
  * Patients suffering from atopic dermatitis: Microparticles are applied to the skin of the forearm both to an area affected by dermatitis and to an area deprived from the disease. A skin biopsy of these two areas is performed.
  The fluorochrome contained in the particle will be detected by confocal microscopy to determine whether the particles have reached beyond the stratum corneum

SECONDARY OUTCOMES:
Assessment of the quantity of fluorescence (assessed by number of pixels on pictures taken with confocal microscopy) | Day 3
  This will be assessed by the number of pixels on pictures taken with confocal microscopy. It will allow for the comparison between patients/healthy volunteers and the comparison of affected/non-affected area in patients

CONTACTS AND LOCATIONS:
Overall Officials: Philippe HUMBERT, Principal Investigator — Centre Hospitalier Universitaire de Besancon
Locations (1):
- Regional University Hospital, Besançon, France